CLINICAL TRIAL: NCT00806650
Title: Development of a Blood Test of Anti-IMP3 Autoantibody and Serum MicroRNA Signature for the Detection of Renal Cell Carcinoma With Metastasis and Metastatic Potential
Brief Title: Anti-IMP3 Autoantibody and MicroRNA Signature Blood Tests in Finding Metastasis in Patients With Localized or Metastatic Kidney Cancer
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07241; CHNMC-07241; CDR0000628796 (Registry Identifier: NCI PDQ); NCI-2015-01327 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gene Expression Profiling; Immunoenzyme Techniques; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Blood draw for diagnosis testing
  Interventions: Genetic: gene expression analysis; Genetic: protein expression analysis; Diagnostic Test: diagnostic laboratory biomarker analysis; Other: immunoenzyme technique; Other: immunohistochemistry staining method

INTERVENTIONS:
Genetic: gene expression analysis — Testing performed on blood draw taken prior to surgery or other treatment and on fresh or frozen primary or metastatic tissue samples
Genetic: protein expression analysis — Testing performed on blood draw taken prior to surgery or other treatment and on fresh or frozen primary or metastatic tissue samples
Diagnostic Test: diagnostic laboratory biomarker analysis — Testing performed on blood draw taken prior to surgery or other treatment and on fresh or frozen primary or metastatic tissue samples
Other: immunoenzyme technique — Testing performed on blood draw taken prior to surgery or other treatment and on fresh or frozen primary or metastatic tissue samples
Other: immunohistochemistry staining method — Testing performed on blood draw taken prior to surgery or other treatment and on fresh or frozen primary or metastatic tissue samples

SUMMARY:
This research trial studies the development of a blood test for detecting anti-insulin-like growth factor II mRNA binding protein 3 (anti-IMP3) antibody and micro ribonucleic acid (microRNA) in patients with renal cell carcinoma (RCC) that has spread to other parts of the body (metastatic) or is limited to the tissue or organ where it began (localized). Anti-IMP3 is a tumor marker that can be detected in many human cancers, including RCC and is likely to be present in the serum (blood) of patients with metastatic or localized RCC. Alterations in microRNA expression has also shown to play a critical role in cancer progression and may be a promising biomarker for patients with RCC. Developing a blood test for anti-IMP3 antibody and microRNA in serum and tissue samples of patients in the laboratory may help doctors find and diagnose RCC earlier, find out how far the disease has spread, and plan effective treatment for RCC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop a blood test by monitoring the titer of IMP3 autoantibody and/or microRNA (miRNA)/small non-coding RNA (snRNA) expression in patients' serum for the early detection of RCC and its recurrence/metastasis.

OUTLINE: Serum samples are collected prior to treatment and analyzed for anti-IMP3 autoantibody titer via enzyme-linked immunosorbent assay (ELISA) and total RNA via sequencing, microarray, and/or quantitative polymerase chain reaction (q-PCR). Previously collected tissue samples are analyzed for IMP3 via immunohistochemistry (IHC).

ELIGIBILITY:
Inclusion Criteria:

Metastatic RCC Patients' Serum Cohort:

* a. Serum samples from patients with metastatic RCC prior to surgical removal of the metastatic and/or primary lesions
* b. Serum samples from patients with localized RCC prior to surgical removal of the lesions
* c. Discarded donors' and patients' discarded/leftover plasma/serum samples from blood bank and other Department of Pathology laboratories
* d. Serum samples from patients with metastatic RCC who had nephrectomies or/and RCC-related biopsies in the referring hospitals

Metastatic RCC Patients' Tissue Cohort:

* Formalin-fixed paraffin-embedded (FFPE) and/or frozen primary and/or metastatic RCC tissue samples from the corresponding patients serum who are included in inclusion criteria (a-b)
* FFPE and/or frozen benign renal tissue samples which are nearby the tumor and remove during surgical procedures from the corresponding patients who are included in inclusion criteria (a-b)
* Discarded/leftover FFPE and frozen renal tissue samples from Department of Anatomic Pathology and its Tumor Bank
* FFPE primary and/or metastatic RCC tissue samples (unstained slides) from the corresponding patients who are included in inclusion criteria (d)

Exclusion Criteria:

Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with metastatic or localized RCC
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2008-07; Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Presence of primary and/or metastatic renal cell carcinoma by IMP3 autoantibody | Baseline
  For the IMP3 autoantibody study, the results of IHC studies of IMP3 on the tissue sections will be used as golden standard to evaluate the sensitivity and specificity of the assay. Statistical significance will be set at P < 0.05 (confidence level of 95%).
Presence of primary and/or metastatic renal cell carcinoma by miRNA/snRNA signature | Baseline
  For the miRNA/snRNA signature study, the patients' clinical presentation of RCC and its recurrence/metastasis will be used as the golden standard to evaluate the sensitivity and specificity of the assay. Statistical significance will be set at P < 0.05 (confidence level of 95%).

CONTACTS AND LOCATIONS:
Overall Officials: Huiqing Wu, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States